CLINICAL TRIAL: NCT01128127
Title: Strategies for Improving Proton Pump Inhibitors (PPIs) Prescription for Gastropathy Prevention Due to Non-steroidal Anti-inflammatory Drugs (NSAIDs) in Primary Health Care
Brief Title: Strategies for Improving Proton Pump Inhibitors (PPIs) Prescription Associated to Non-steroidal Anti-inflammatory Drugs (NSAIDs)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: Fundación Canaria de Investigación y Salud (Other Government)
Responsible Party: Dr. Pedro Serrano-Aguilar, Servicio de Evaluación. Servicio Canario de Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PI 43 08
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Adverse Events
Keywords: knowledge translation; prescription; primary care; NSAID; PPI; Gastrointestinal damage; Inappropriate prescription

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multifaceted intervention 1 (Experimental): psycho-educational workshop + audit-feedback + computer-based clinical decision support system (CCDSS) + usual intervention
  Interventions: Behavioral: Group education, audit-feedback and computer support
- Multifaceted intervention 2 (Experimental): audit-feedback + computer-based clinical decision support system (CCDSS) + usual intervention
  Interventions: Behavioral: Audit-feedback and computer support
- Control (Active Comparator): usual intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Group education, audit-feedback and computer support — Psycho-educational group workshop: two theory-practice sessions on both evidence-based guidelines on PPI-NSAID prescription and communication and negotiation skills to deal with patients. All participants will fill out an initial questionnaire concerning prescribing patterns and barriers to appropriate prescription. All attendees will be given a reminder printed material designed to give the necessary information in a brief fashion and for maximal visual impact.
  Audit-Feedback: participants will receive, monthly and by e-mail, an individualized report with data of their own appropriate/inappropriate PPI prescriptions and avoidable costs.
  CCDSS: interactive computer program designed to assist physicians with decision making when prescribing PPI associated to NSAID. It consists in pop-up alert screens that aim to influence prescription choice according to each patient characteristics and evidence-based clinical guidelines.
  Arms: Multifaceted intervention 1
Behavioral: Audit-feedback and computer support — Audit-Feedback: participants will receive, monthly and by e-mail, an individualized report with data of their own appropriate/inappropriate PPI prescriptions and avoidable costs
  CCDSS: interactive computer program designed to assist physicians with decision making when prescribing PPI associated to NSAID. It consists in pop-up alert screens that aim to influence prescription choice according to each patient characteristics and evidence-based clinical guidelines.
  Arms: Multifaceted intervention 2
Behavioral: Control — Usual intervention includes:
  Compulsory attendance both to courses (10-12 hours) and to short sessions (around 30 min.) on the rational use of drugs held in groups and during working hours. Each primary care physician attends to 1-2 courses and 3-4 short sessions per year.
  Every three months, physicians receive a feedback paper with information on his/her own prescribing overall costs comparing to his/her primary care center average cost.
  Distribution of a printed booklet of recommendations, delivered personally or through mass mailings, on the prescribing of PPI-NSAID.
  Arms: Control

SUMMARY:
Background

Despite the low prevalence of serious complications associated with non-steroidal anti-inflammatory drugs (NSAIDs) use, there is a widespread use of gastroprotective proton pump inhibitors (PPIs) in order to prevent adverse effects. Inappropriate prescribing of PPIs includes overprescribing for inappropriate indications and the misuse of first choice in their class in terms of efficacy, safety and cost. A series of recommendations, based on the best available scientific evidence, has been established to justify prophylaxis with PPIs associated to NSAIDs. Therefore, there is the need to encourage the incorporation of this knowledge to guide decisions of physicians with the objective of improving patient health and sustainability of the Public Health Service. Although since long ago there is a great concern regarding rational use of drugs, the available evidence for the most appropriate strategies to improve prescribing is scarce. Passive dissemination of research findings are generally ineffective and at best result in small changes in practice. Multifaceted intervention targeting different barriers to change are more likely to be effective than single intervention.

Objectives

The objective of this study is to evaluate the effectiveness of two educational multifaceted strategies aimed at improving PPIs prescription associated to NSAIDs use in primary care. We will also compare the cost-effectiveness of such strategies.

Hypothesis

It is hypothesized that a quality improvement intervention directed to primary care physicians will decrease inappropriate PPIs prescriptions associated to NSAIDs prescription.

Methodology

A three-arm prospective quasi-randomized controlled trial will test the effectiveness of two strategies for improving PPI prescription associated to NSAID in primary care context. Three of the Canary Islands will be selected and randomized to either a experimental multifaceted intervention (group education+audit-feedback+CCDSS) group, a experimental multifaceted intervention (audit-feedback+CCDSS) group, or a control group (usual intervention). From each of these islands, 6-8 primary care centers will be randomly selected to received the intervention practices. All family physicians working at each randomly selected primary care center were mandatorily included. Primary outcome measure is reduction of inappropriate PPI prescription. The efficacy of the intervention will be examined within a 3, 6 and a 12 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians

Exclusion Criteria:

* Participating as a subject in any other clinical research study
* Have received any other intervention on the subject within the last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Rate of inappropriate PPI prescriptions | one year
  Change in the proportion of inappropriate PPI prescription associated with NSAID prescription

CONTACTS AND LOCATIONS:
Overall Officials: Pedro G Serrano-Aguilar, MD, PhD, Principal Investigator — Servicio de Evaluación. Servicio Canario de Salud; Yolanda Ramallo-Fariña, BSc Statist, Study Chair — Fundación Canaria de Investigación y Salud; Maria M Trujillo-Martín, PhD, Study Chair — Fundación Canaria de Investigación y Salud; Melany Worbes-Cerezo, BAEcon, Study Chair — CIBER Epidemiología y Salud Pública (CIBERESP), Spain; Renata Linertova, BA Econ, Study Chair — Fundación Canaria de Investigación y Salud; Francisco J Hernández-Diaz, MD, PhD, Study Chair — Servicio Canario de Salud; Miguel A Hernández-Rodríguez, MD, PhD, Study Chair — Servicio Canario de Salud; Pedro Gonzalez-Leandro, PhD, Study Chair — University of La Laguna; Livia García-Pérez, PhD, Study Chair — University of La Laguna
Locations (1):
- Servicio de Evaluación. Servicio Canario de Salud, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain